CLINICAL TRIAL: NCT04169399
Title: Toripalimab Plus Stereotactic Body Radiotherapy for Hepatocellular Carcinoma With Portal Vein Tumor Thrombus: a Single-arm, Prospective Trial
Brief Title: Toripalimab Plus Stereotactic Body Radiotherapy for HCC With PVTT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S1001
Record Dates: First submitted 2019-11-17; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Toripalimab; Stereotactic body radiotherapy; Portal vein tumor thrombus
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — toripalimab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab plus SBRT (Experimental): Participants received 240mg toripalimab intravenously every 3 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent. Participants recevied Stereotactic body radiotherapy. Radiotherapy dose was 36 ~ 54Gy, divided into 6 times of irradiation, and the radiation was performed within 2 weeks.
  Interventions: Drug: Toripalimab; Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Drug: Toripalimab — 240mg intravenously every 3 weeks
Radiation: Stereotactic body radiotherapy — Radiotherapy dose was 36 ~ 54Gy, divided into 6 times of irradiation, and the radiation was performed within 2 weeks.

SUMMARY:
To explore the efficacy and safety of toripalimab plus stereotactic body radiotherapy for hepatocellular carcinom with portal vein tumor thrombus.

DETAILED DESCRIPTION:
Programmed Cell Death Protein-1 (PD-1) was effective and tolerable in patients with advanced hepatocellular carcinoma. Additionally, previous studies showed that stereotactic body radiotherapy (SBRT) was effective for hepatocellular carcinoma with portal vein tumor thrombus (PVTT). No study has evaluated the efficacy and safety of toripalimab plus SBRT for hepatocellular carcinoma with PVTT. Thus, the investigators carried out this prospective study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to mRECIST criteria
* The normal liver volume in the non-target area was greater than 700ml
* Portal vein tumor thrumbus confirmed in two image techniques
* Eastern Cooperative Oncology Group performance status of 0 to 2
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* With no previous radiotherapy and immunotherapy
* Not applicable for transarterial chemoembolization, surgical resection, and local ablative therapy.
* The following laboratory parameters:

Platelet count ≥ 75,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/ L Serum albumin ≥ 30 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3 Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-17 (Actual); Primary Completion 2020-11-17 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 6 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on iRECIST, or date of death, whichever occurred first

SECONDARY OUTCOMES:
Overall survival (OS) | 6 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.
Objective Response Rate (ORR) | 6 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on iRECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions.
Adverse Events | 6 months
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China